CLINICAL TRIAL: NCT01468493
Title: A Prospective Controlled Follow-up of Serum Soluble Urokinase Receptor in the Cyclosporine A-treated Patients With Steroid-dependent and Steroid-resistant Focal Segmental Glomerulosclerosis
Brief Title: A Prospective Controlled Study of Serum suPAR in the CsA-treated FSGS Patients
Acronym: SuparSDRF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Wei Shi, Director of renal division of Guangdong General Hospital, Guangdong Provincial People's Hospital
Other Study IDs: GGH-1-1
Record Dates: First submitted 2011-10-29; First posted 2011-11-09 (Estimated); Last update posted 2017-04-24 (Actual); Status verified 2017-04

CONDITIONS: FSGS
Keywords: FSGS; suPAR

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- steroid-sensitive FSGS
- steroid-dependent and resistant FSGS
- Healthy volunteers

SUMMARY:
The purpose of this study is to determine whether the improved responsiveness to treatment achieved by CsA in patients with steroid-resistant or steroid-dependent FSGS could be explained by CsA's inhibitory action on the circulating suPAR expression.

ELIGIBILITY:
Inclusion Criteria:

* Age at entry is between 14 and 70 years
* biopsy-proven primary FSGS
* proteinuria >=3 g/day
* without corticosteroids or CsA treatment before entry

Exclusion Criteria:

* Chronic Inflammatory Diseases
* malignant tumor
* diabetes mellitus
* contraindications for the treatment of corticosteroids or CsA treatment
* untolerate to or unwilling to accept corticosteroids or CsA treatment

Ages: 14 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 1)the patients with steroid-sensitive FSGS;2)the cyclosporine A-treated patients with steroid-dependent and steroid-resistant FSGS;3)the healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2011-01; Primary Completion 2019-01 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
serum suPAR level when proteinuria reduction >=50% or complete remission | 6 months after steriod alone or CsA plus steriod treatment
  serum suPAR level when proteinuria reduction of >=50% or complete remission occurs within <=6 months of steroid alone or CsA plus steroid treatment

SECONDARY OUTCOMES:
serum suPAR level after 6 months of steroid or CsA treatment without remission | 6 months after steroid alone or CsA plus steroid treatment
  serum suPAR level after 6 months of steroid alone or CsA plus steroid treatment without remission

CONTACTS AND LOCATIONS:
Overall Officials: Wei Shi, MD,PhD, Principal Investigator — Nephrology Dept.,Guangdong General Hospital
Locations (1):
- Nephrology Dept.,Guangdong General Hospital, Guangzhou, Guangdong, China